CLINICAL TRIAL: NCT03932903
Title: Using Real Time Mobile Health Approaches to Understand and Promote Oral Chemotherapy Adherence in Adolescents and Young Adults With Leukemia
Brief Title: Mobile Health Intervention to Support Oral Chemotherapy Adherence in Adolescents and Young Adults With Leukemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Alex Psihogios, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 19-016325
Record Dates: First submitted 2019-04-24; First posted 2019-05-01 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma
Keywords: Adherence; Adolescent; Young Adult; Mobile Health; Oncology
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms

STUDY DESIGN:
Intervention Model Description: This study involve a 28-day micro-randomized pilot trial (i.e., a sequential factorial design) of a just-in-time adaptive intervention called ADAPTS ADAPTS is an app that will deliver contextually-tailored mobile messages (adapted to current states, such as mood, pain, and location) designed to promote oral chemotherapy adherence. Each AYA in the study (planned n=30) will be micro-randomized (with a 60% probability) to receive a contextually-tailored message each day that supports abilities to self-manage and maintain adherence, delivered prior to their scheduled dose, over a 28-day period (i.e., the period between follow-up appointments). The remaining 40% of days, participants will be assigned to receive no messages (i.e., no intervention).
  We will also request, but not require, that a caregiver enrolls in the study and pilots the caregiver version of the app (planned n=30 caregivers). The caregiver app does not include any micro-randomization.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contextually-tailored Mobile Messages for Adherence (Experimental): AYA participants will be micro-randomized to receive contextually-tailored mobile messages designed to promote their oral chemotherapy adherence, with a 60% probability of receiving a contextually-tailored message each day.
  Interventions: Behavioral: ADAPTS (ADherence Assessments and Personalized Timely Support).
- No messages (No Intervention): All participants will also be micro-randomized to not receive messages on some days of the intervention (~40% of the time).

INTERVENTIONS:
Behavioral: ADAPTS (ADherence Assessments and Personalized Timely Support). — ADAPTS is a mobile app intervention that integrates contextually-tailored mobile messages and decision rules about when to deliver the messages, with the ultimate goal of improving oral chemotherapy adherence in AYAs with acute lymphoblastic leukemia and lymphoma. AYA participants will be micro-randomized to receive messages on some days that are adapted to their current characteristics (e.g., mood, pain, location) and designed to promote adherence, and no messages (no intervention) on other days. Other features in the app include a medication calendar that syncs with the electronic medication monitor (eCAP) to track daily adherence. A caregiver version of ADAPTS is also available, providing daily surveys (but no randomized mobile messages) and the medication calendar so that dyads can mutually track adherence.
  Arms: Contextually-tailored Mobile Messages for Adherence

SUMMARY:
This is a small-scale micro-randomized clinical trial of a new mobile just-in-time adaptive intervention (JITAI) designed to promote oral chemotherapy adherence in adolescents and young adults (AYA) with acute lymphoblastic leukemia (ALL). The goals of this study are to determine intervention feasibility and acceptability.

DETAILED DESCRIPTION:
This is two-month study involving a 28-day run-in period (no intervention), followed by a 28-day micro-randomized pilot trial (i.e., a sequential factorial design) of a just-in-time adaptive intervention (JITAI) called ADAPTS (ADherence Assessments and Personalized Timely Support). ADAPTS is an app that integrates contextually-tailored mobile messages designed to promote adherence to an oral chemotherapy called 6-mercaptopurine (6-MP). Participants in the study will electronically-monitor 6-MP adherence with eCAPs for 28 days (approximately one month to establish baseline adherence before introducing the intervention). On approximately Day 29, they will download and use the app while continuing to monitor their adherence for the next 28 days. ADAPTS is an app that is available for Android and Apple devices, and has an Adolescent/Young Adult (AYA) version (i.e., the primary user) and a Caregiver version. ADAPTS delivers ecological momentary assessment (EMA) surveys each afternoon to AYAs and caregivers, at the same time prior to the evening 6-MP dose, for the 28-day period. Based on EMA responses, ADAPTS sends contextually-tailored mobile messages to AYAs (e.g., based on self-reported fatigue, mood) and objective data (e.g., weekend vs. weekday). After receiving a contextually-tailored message, AYAs will be asked to acknowledge receipt of the message by pressing a "thumbs up" or "thumbs down" button, to indicate whether or not they liked the message, or a "snooze" button indicating that it was not a good time to receive the message. Some features in ADAPTS are designed for AYAs and their caregivers to use together, such as a medication calendar that syncs with the eCAP and can be viewed by both members of the dyad. Following the 28-day intervention period, eCAPS will be returned and downloaded during the clinic appointment. AYAs and caregivers will complete a brief acceptability survey electronically via REDCAP, rating ADAPTS on a 5-point Likert scale to assess satisfaction, perceived appropriateness, perceive positive effects, perceived demands, and potential for future use. Exit interviews will also be conducted, audio-recorded, and transcribed to further assess acceptability. For feasibility, the following variables will be tracked: (1) screening rates, (2) recruitment rates, (3) % acknowledged micro-randomized messages, (4) technical difficulties (e.g., micro-randomized messages received when intended), (5) retention rates, and (6) completed assessments (EMA, eCAPS, post-measures).

ELIGIBILITY:
AYA Inclusion Criteria:

* Ages 14-29
* Diagnosed with acute lymphoblastic leukemia (ALL) or lymphoma
* In the maintenance phase, completed at least one cycle and has at least one month of maintenance therapy remaining.
* Prescribed 6-mercaptopurine (6MP)
* English language proficiency
* For AYA <18, must have informed consent from their caregiver.

AYA Exclusion Criteria:

* Cognitive impairments that would limit ability to complete measures, determined by the medical team
* Absence of inclusion criteria above.

Caregiver Inclusion Criteria:

* Nominated by the AYA as a primary caregiver involved in cancer care (can be a parent, relative, partner, friend)
* English language proficiency

Caregiver Exclusion Criteria:

- Absence of inclusion criteria above.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Technical Difficulties | 28-day intervention period
  Number of technical glitches and errors experienced in implementing the intervention
Retention Rate | Up to 12 months
  Number of AYA (and caregiver) subjects who complete the intervention, out of the total number of subjects enrolled in the study (target of 75% or more)
Screening Rate | Up to 12 months
  Number of AYA patients (and matched caregivers) referred and screened for the study
Intervention Engagement | 28-day intervention period
  Number of 1) viewed and 2) acknowledged micro-randomized text messages
Recruitment Rate | Up to 12 months
  Number of AYA patients (and matched caregivers) enrolled in the study out of those who were eligible and invited to participate (target of 75% or more)
Intervention Acceptability | At completion of 28-day intervention period
  5-point numerical Likert scale; ranging from 0 (not at all) to 4 (completely) to rate intervention acceptability (including satisfaction, appropriateness, perceived positive effects, potential for future use).

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra M Psihogios, Ph.D., Principal Investigator — Northwestern University
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhatia S, Landier W, Hageman L, Kim H, Chen Y, Crews KR, Evans WE, Bostrom B, Casillas J, Dickens DS, Maloney KW, Neglia JP, Ravindranath Y, Ritchey AK, Wong FL, Relling MV. 6MP adherence in a multiracial cohort of children with acute lymphoblastic leukemia: a Children's Oncology Group study. Blood. 2014 Oct 9;124(15):2345-53. doi: 10.1182/blood-2014-01-552166. Epub 2014 May 14. PMID 24829202
- [Background] Modi AC, Pai AL, Hommel KA, Hood KK, Cortina S, Hilliard ME, Guilfoyle SM, Gray WN, Drotar D. Pediatric self-management: a framework for research, practice, and policy. Pediatrics. 2012 Feb;129(2):e473-85. doi: 10.1542/peds.2011-1635. Epub 2012 Jan 4. PMID 22218838
- [Background] Klasnja P, Hekler EB, Shiffman S, Boruvka A, Almirall D, Tewari A, Murphy SA. Microrandomized trials: An experimental design for developing just-in-time adaptive interventions. Health Psychol. 2015 Dec;34S(0):1220-8. doi: 10.1037/hea0000305. PMID 26651463
- [Background] Nahum-Shani I, Smith SN, Spring BJ, Collins LM, Witkiewitz K, Tewari A, Murphy SA. Just-in-Time Adaptive Interventions (JITAIs) in Mobile Health: Key Components and Design Principles for Ongoing Health Behavior Support. Ann Behav Med. 2018 May 18;52(6):446-462. doi: 10.1007/s12160-016-9830-8. PMID 27663578
- [Background] Psihogios AM, Li Y, Butler E, Hamilton J, Daniel LC, Barakat LP, Bonafide CP, Schwartz LA. Text Message Responsivity in a 2-Way Short Message Service Pilot Intervention With Adolescent and Young Adult Survivors of Cancer. JMIR Mhealth Uhealth. 2019 Apr 18;7(4):e12547. doi: 10.2196/12547. PMID 30998225
- [Background] Psihogios AM, Fellmeth H, Schwartz LA, Barakat LP. Family Functioning and Medical Adherence Across Children and Adolescents With Chronic Health Conditions: A Meta-Analysis. J Pediatr Psychol. 2019 Jan 1;44(1):84-97. doi: 10.1093/jpepsy/jsy044. PMID 29982694
- [Background] McGrady ME, Brown GA, Pai AL. Medication adherence decision-making among adolescents and young adults with cancer. Eur J Oncol Nurs. 2016 Feb;20:207-14. doi: 10.1016/j.ejon.2015.08.007. Epub 2015 Sep 12. PMID 26372619
- [Background] Butow P, Palmer S, Pai A, Goodenough B, Luckett T, King M. Review of adherence-related issues in adolescents and young adults with cancer. J Clin Oncol. 2010 Nov 10;28(32):4800-9. doi: 10.1200/JCO.2009.22.2802. Epub 2010 Mar 8. PMID 20212260